CLINICAL TRIAL: NCT05353790
Title: Macro- and Micro- Vascular Function and Related Cognitive Effects in Response to Dietary Exchanges With Avocado and Mango in Pre-diabetes.
Brief Title: Dietary Exchanges With Avocado and Mango in Pre-diabetes
Acronym: AVMa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Hass Avocado Board (Other); National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2021-67
Record Dates: First submitted 2022-02-20; First posted 2022-04-29 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pre Diabetes; Vascular Stiffness; Vascular Dilation; Cognitive Change; Retinal Vascular
MeSH Terms: conditions — Glucose Intolerance | interventions — Meals

STUDY DESIGN:
Who Masked: Participant
Masking Description: Four one-week meal plans for each Active and Control intervention will be developed and given twice in random order to allow for a partially controlled dietary regimen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avocado mango meal plan (Experimental): 2 meals and snacks per day, including 1 avocado + 1 cup of mango, covering 75% of daily calories needs,
  Interventions: Other: Meals + snacks: Avocado mango
- Control meal plan (Other): 2 meals and snacks per day, without avocado and mango, covering 75% of daily calories needs
  Interventions: Other: Meals + snacks: control

INTERVENTIONS:
Other: Meals + snacks: control — 8 weeks meal plans matched in calories (but not macronutrients or fiber) equivalent to 1 avocado + 1 cup of mango per day
  Arms: Control meal plan
Other: Meals + snacks: Avocado mango — 8 weeks meal plans provide1 avocado + 1 cup of mango per day
  Arms: Avocado mango meal plan

SUMMARY:
The research is designed as a randomized, 2-arm, parallel, controlled, human clinical trial to investigate the effects of avocado and mango consumption for 8 weeks on indices of macro- and micro- vascular function in individuals with prediabetes. FMD of the brachial artery, pulse wave velocity (PWV), central blood pressure (cBP), and Optical Coherence Tomography Angiography (OCTA) of the eye will be used for vascular assessments. The research plan will also explore cognitive and kidney function benefits of regular avocado and mango intake using specified cognitive tasks and kidney function biomarkers

DETAILED DESCRIPTION:
Recruited subjects must meet all eligibility criteria, sign and date a written Institutional Review Board (IRB)-approved Informed Consent Form.

The trial will test 2 dietary conditions which will be fresh fruit (1 avocado and 1 mango) compared to a control arm matched in calories (but not macronutrients or fiber) equivalent to 1 fresh Hass avocado + 1 cup of mango per day. Participants will be given general meal plans, including specific foods assnacks or meals to include in their diet daily.

* Pre-Screening To learn more about the study and to pre-qualify, potential subjects can call the CNRC or visit the website posted on recruitment flyers or from other recruitment materials. If they call the CNRC, a staff member will provide a brief background on the study and ask a series of questions from a pre-screening questionnaire to see if they may be eligible to participate. The same questionnaire is available on the website and can be filled out by potential subjects online. The pre-screening questionnaire includes self-reported information about health status and lifestyle factors that can be used to determine if someone is not eligible for the study.
* Information Session and Screening Session Information Session and Screening Visit may occur simultaneously or Information Session may occur prior to Screening Visit. Prior to the Screening Visit, potential subjects will be asked to arrive at the CNRC after an overnight-fast (stop eating after 10 pm) and be well-hydrated. Subjects should aim for drinking at least 8-10 cups of water the 24 h prior to the Screening Visit.

Information Session: At the CNRC, pre-screened subjects will participate in an Information Session where they will be informed of all study procedures and study schedules. If willing to adhere to all study procedures and schedules, they will be asked to read, ask questions, signand date the Institutional Review Board (IRB) approved Informed Consent Form (ICF) before any laboratory or study screening procedures begin.

Screening Visit: After meeting eligibility criteria for blood glucose (BG) and blood pressure (BP) measures, subjects will advance to further screening procedures which will include a comprehensive chemistry panel plus TSH, anthropometric measurements (height, weight, waist circumference, body composition), BMI (calculated from height and weight), medical history, prior and concomitant medication, and dietary supplements use, and completion of a series of questionnaires relating to their general health and lifestyle.

After confirming eligibility through blood test results, subjects will then be scheduled for a visit to the Illinois Eye Institute (IEI) for a screening eye exam. During this exam, drops to check the eye pressure and drops to dilate eyes will be used. Based on study eligibility criteria subjects may be invited to participate in the study. A Pre-Study Visit and all Test Day Visits will be scheduled before leaving the CNRC or shortly thereafter.

-Pre-Study Visit, Randomization, and Cognitive assessment The pre-study visit is for training on various aspects of the study. In addition, subjects will be randomized for more specific study protocol information (eg., dietary inclusion of study foods). The Pre-Study Visit will also include a baseline cognitive function test. This will include visiting instructions for preparing for the cognitive test (eg., fasting instructions, waiting to eat breakfast and having morning coffee/tea at the clinic, etc). Each subject will come to the CNRC in fasting (10 hours) state for one pre-scheduled Pre-Study Visit, where they will receive a breakfast meal to consume onsite and complete the baseline cognitive testing and then proceed to instructions on the process for completing various aspects of the research protocol, including but not limited to, the online 24 h dietary recalls (via ASA24 program), weekly visits for food pick up, incorporating foods into diet, plan for eye exams, and more. They will also be provided with all study instructions for fasting before each major test day, completing check-off diaries to help with study compliance, text/email verification receiving appointment reminders, etc.

Test Day Visits: All subjects will report to the CNRC on a weekly basis unless conditions outside our control require less frequent person-to-person interaction. In this case, however, alternatives mechanisms will be instituted to ensure contact with subjects and delivery of the product. Visit 1, Visit 5, and Visit 9 will have two phases (a visit at IEI & b visit at CNRC). specifically, subjects will go to the IEI for collection of the OCT-A images (Visit 1a, 5a, and 9a) 1-5 days prior to the visit at CNRC. Visits at CNRC: Visit 1b, Visit 5b, and Visit 9b encompass all study procedures (except for the cognitive battery, which is performed at Pre-Study and Visit 8). A fasting blood sample, FMD, PWV, cBP, anthropometrics, and 24 h recall will all be assessed. Subjects will be given a standardized breakfast and the FMD repeated 1.5 h later. Thereafter, subject will be given groceries and study-specific food products and reminded how to include in their diet. A Test Day Visit Questionnaire to report compliance with study instructions (after first visit), dietary tolerance and general health status (any illnesses in the 7 days before the Test Day Visit), change in meds, will be given/collected. To minimize vascular and metabolic variability due to hormone fluctuations associated with the menstrual cycle women will be studied in the follicular phase of their menstrual cycle. The 8-week intervention allows for scheduling individuals' females accordingly. For subjects willing to return 2 months after discontinuing treatment, Visit 9 will be repeated for follow-up. This visit will not be considered part of "completer" analysis but will provide insight for research and study designs. Blood Donation Guidelines indicated that for each subject no more than 550 mL of blood be collected in a 56-day period. The amount of blood collected in this study will be far below donation guidelines (~70 mL) over the course of the study.

-Food pick up days (CNRC, IllinoisTech) Bodyweight, compliance records, general health questionnaire, and dietary tolerance questionnaire will be completed. Food provided per randomization.

Meal plans. Four one-week meal plans for each Active and Control intervention will be developed and given twice in random order to allow for a partially controlled dietary regimen.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 25-70 year- Fasting blood glucose concentration between 100 mg/dL and 125 mg/dL at screening visit
* Blood pressure 120-160 mmHg systolic or 80-100 mm/Hg diastolic at screening visit
* Nonsmokers (past smokers can be allowed if they have abstinence for minimum of 12 months)
* Judged to be in good health on the basis of the medical history (i.e., no clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications that would interfere with outcomes of the study, (e.g., lipid lowering medications, anti-inflammatory drugs, dietary supplements, etc.)
* Able to provide informed consent
* Able to comply and perform the procedures requested by the protocol (follow the dietary plans, come to scheduled visits, record food intake in a diary, complete questionnaires, provide blood samples and complete other tests (eye and brain/cognitive function)
* Able to maintain usual physical activity pattern
* Able to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during study visit

Exclusion Criteria:

* Men and women who have blood pressure >160 mmHg (systolic)/100 mmHg (diastolic) at screening visit
* Men and women who have fasting blood glucose concentration <100 or >125 mg/dL at screening visit
* Abnormal Thyroid-stimulating Hormone (TSH) at screening visit
* Men and women with diabetes
* History of cardiovascular event, respiratory, renal, gastrointestinal, hepatic or eye disease or surgery (e.g., heart failure, myocardial infarction, stroke, angina, related surgeries, etc.) that, in the opinion of the investigator, could interfere with the interpretation of the study results.
* High refractive error (+/- 6.00 D, axial length greater than 26 mm or less than 22mm), astigmatism >3.00D, impaired vision/not correctible to 20/20, high eye pressures (>21 mmHg) and narrow angles (< grade 3 Van Herick) in the study eye as confirmed by screening eye exam at IEI screening visit
* Head injury in past 6 months
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Taking medication or dietary supplements that may interfere with the outcomes of the study, (e.g., antioxidant supplement, anti-inflammation, lipid-lowering medication, blood pressure-lowering medication, etc.). Subjects may choose to go off dietary supplements (requires 30-day washout; e.g., fish oil, etc.)
* Vegan or other extreme dietary regimens (e.g., Atkins diet, etc.) as judged by the investigator
* Known or suspected intolerance, allergies or hypersensitivity to study foods or treatments
* Current smoker or smoked/vaped within the last 12 months
* Unstable weight: Actively losing or gaining weight or trying to lose or gain weight. Gained or lost weight +/- 5 kg (11 lbs.) in previous 2 months.
* Substance (alcohol or drug) abuse within the last 2 years
* Present with significant psychiatric or neurological disturbances
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are lactating
* Major trauma or a surgical event within 2 months or longer depending on trauma or event and after consultation with PI.
* Has used antibiotics within the previous 2 months
* History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional
* Excessive coffee and tea consumers (> 4 cups/d)
* Donated blood within last 3 months
* Men and women who do excessive exercise regularly or are an athlete
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months
* Unusual working hours (e.g., working overnight; 3rd shift)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in vascular function measured by Flow-mediated vasodilation of brachial artery | baseline-8 weeks
  Macro-vascular assessment by Ultrasonography
Changes in Pulse Wave Velocity | baseline-8 weeks
  fasting state, Macro-vascular assessment by SphygmaCor technology:
Changes in Central Blood pressure | baseline-8 weeks
  fasting state, Macro-vascular assessment by SphygmaCor technology:
Changes in plasma biomarkers:fasting glucose | baseline-8 weeks
  Randox automated clinical analyzer
Changes in plasma biomarkers: fasting insulin | baseline-8 weeks
  Randox automated clinical analyzer
Changes in plasma biomarkers:lipid profile | baseline-8 weeks
  Randox automated clinical analyzer, total cholesterol,LDL cholesterol, HDL cholesterol, triglycerides
Changes in plasma biomarkers and measures of inflammation concentration: IL-6 | baseline-8 weeks
  IL-6 (ELISA, RnD systems)
Changes in plasma biomarkers and measures of inflammation concentration: ICAM | baseline-8 weeks
  ICAM (ELISA, RnD systems)
Changes in plasma biomarkers and measures of inflammation concentration: VCAM | baseline-8 weeks
  VCAM (ELISA, RnD systems)
Changes in plasma biomarkers and measures of brain-derived neurotrophic factor: BDNF | baseline-8 weeks
  BDNF (ELISA, RnD systems)
Changes in plasma biomarkers and measures of brain-derived neurotrophic factor: IGF1 | baseline-8 weeks
  IGF1 (ELISA, RnD systems)
Changes in Kidney function markers | baseline-8 weeks
  serum creatinine

SECONDARY OUTCOMES:
Changes in Foveal Avascular Zone area | baseline-8 weeks
  Microvascular assessment by OCT-A
Changes in Vascular Density superficial and deep | baseline-8 weeks
  Microvascular assessment by OCT-A
Changes in Vascular branch number | baseline-8 weeks
  Microvascular assessment by OCT-A
Changes in Cognitive Function | baseline-8 weeks
  Wide Range Achievement Test-4th Edition, Reading Subtest (WRAT-4 Reading)
Changes in Cognitive Function-1 | baseline-8 weeks
  California Verbal Learning Test-2nd Edition (CVLT-II), including short and long delays
Changes in Cognitive Function-2 | baseline-8 weeks
  Wechsler Adult Intelligence Scale-4th Edition, Matrix Reasoning subset (WAIS-IV MR
Changes in Cognitive Function-3 | baseline-8 weeks
  Trail Making Test A & B
Changes in Cognitive Function-4 | baseline-8 weeks
  WAIS-IV Digit Span subtest (DS)
Changes in Cognitive Function-5 | baseline-8 weeks
  Stroop
Changes in Cognitive Function-6 | baseline-8 weeks
  Verbal Fluency Task (FAS & Animals)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No